## **Statistical Analysis Plan**

Clinical Trial Protocol EMR200505\_506

Identification No.

**Title** An interventional, pilot study to evaluate the efficacy

of oral nicorandil on improving microvascular function in female non - obstructive CAD patients

(SPET study)

Trial Phase IV

Investigational Medicinal Nicorandil (SIGMART® Tablets 5.0 mg) / Oral / t.i.d,

**Product** 12 weeks

Clinical Trial Protocol Protocol Amendment <III> / 15 Apr 2018

Version

Statistical Analysis Plan Author PPD , Study Statistician

Statistical Analysis Plan 13FEB2019 / Version 2.0

**Date and Version** 

Statistical Analysis Plan Reviewers <u>MakroCare</u>

1. PPD

2. PPD

Merck Serono

1. PPD

This document is the property of Merck KGaA, Darmstadt, Germany, or one of its affiliated companies.

It is intended for restricted use only and may not – in full or part – be passed on, reproduced, published or used without express permission of Merck KgaA, Darmstadt, Germany or its affiliate.

Copyright © 2019 by Merck KgaA, Darmstadt, Germany or its affiliate. All rights reserved.



# 1. Signature Page

Statistical Analysis Plan: EMR200505\_506

An interventional, pilot study to evaluate the efficacy of oral nicorandil on improving microvascular function in female non – obstructive CAD patients (SPET study)

| PPD | PPD |
|-----------------------|-------------------|
| Signature | Date of Signature |
| Trial Biostatistician | |
| PPD | |
| TIL PPD | |
| Tel.: PPD | 2.1 |
| Email: PPD | |



| 2. | Table of Contents |
|---|---|
| 1. | Signature Page2 |
| 2. | Table of Contents3 |
| 3. | List of Abbreviations and Definition of Terms5 |
| 4. | Modification History7 |
| 5. | Purpose of the Statistical Analysis Plan8 |
| 6. | Summary of Clinical Trial Features9 |
| 7. | Sample Size16 |
| 8. | Overview of Planned Analyses16 |
| 9. | Changes to the Planned Analyses in the Observational Study Protocol |
| 10. | Analysis Sets16 |
| 11. | General Specifications for Statistical Analyses17 |
| 12. | Trial Subjects18 |
| 12.1 | Disposition of Subjects and Discontinuations18 |
| 12.2 | Outliers19 |
| 13. | Demographics and Other Baseline Characteristics19 |
| 13.1 | Demographics |
| 13.2 | Medical History20 |
| 14. | Previous or Concomitant Medications/Procedures |
| 15. | Treatment Compliance and Exposure |
| 16. | Endpoint Evaluation |
| 16.1 | Primary Endpoint Analyses |
| 16.2 | Secondary Endpoint Analyses |
| 17. | Safety Evaluation |
| 17.1 | Adverse Reactions / Events |
| 17.1.1 | All Adverse Events |
| 17.1.2 | Adverse Events Leading to Trial or Treatment Discontinuation25 |
| 17.2 | Deaths, Other Serious Adverse Events, and Other Significant Adverse Events |
| 17.2.1 | Deaths25 |
| 17.2.2 | Serious Adverse Events |
| 17.3 | Clinical Laboratory Evaluation |



| Nicorandil<br>EMR200505_50 | 6 | Version 2.0, 13FEB2019 |
|---|---|---|
| 17.4 | Electrocardiogram (ECG): | 28 |
| 17.5 | Vital Signs | 29 |
| 17.6 | Physical Examination | 29 |
| 18. | Benefit risk assessment | 30 |
| 19. | References | 30 |
| 20. | Appendices | 30 |



## 3. List of Abbreviations and Definition of Terms

ACEI Angiotensin-Converting Enzyme Inhibitor(s)

AE Adverse Event

ALT Alanine Transaminase

ARB Angiotensin II Receptor Blockers

AST Aspartate Aminotransferase

BUN Blood Urea Nitrogen

CAD Coronary Artery Disease

CCB Calcium Channel Blocker

CFR Coronary Flow Reserve

CI Confidence Intervals

CKMB Myocardial Enzymes

CMD Coronary Microvascular Dysfunction

CREAT Creatinine

CRF Case Report Form

CTR Clinical Trial Report

DBP Diastolic Blood Pressure

ECG Electrocardiogram

EF Ejection Fraction

HDL High Density Lipoprotein

ICF Informed Consent Form

ICH International Conference on Harmonization

ITT Intention to Treat

IVST Interventricular Septum Thickness



K<sub>ATP</sub> Potassium

LDL Low Density Lipoprotein

LVESD Left Ventricular End Systolic Diameter

MedDRA Medical Dictionary for Regulatory Activities

MBF Myocardial Blood Flow

MFR Myocardial Blood Flow Reserve

MPR Medication Possession Ratio

NYHA New York Heart Association

PET Positron Emission Tomography

PP Per Protocol

PT Preferred Term

PWT Posterior Wall Thickness

SAE Serious Adverse Event

SAP Statistical Analysis Plan

SAQ Seattle Angina Questionnaire

SAS Statistical Analysis System

SBP Systolic Blood pressure

SEM Standard Error of Mean

SOC System Organ Class

TEAE Treatment Emergent Adverse Events

UCG Ultrasound Cardiogram

VOC Voltage-sensitive Calcium Channels



# 4. Modification History

| Unique Identifier<br>for SAP Version | Date of SAP<br>Version | Author | Changes from the Previous<br>Version |
|---|---|---|---|
| 0.1 | 23 DEC 2016 | PPD | Baseline Version |
| 1.0 | 11 APR 2017 | PPD | Final Version |
| 1.1 | 27 SEP 2018 | PPD | Based on the amended protocol and CRF |
| 1.2 | 16 OCT 2018 | PPD | Based on client comments |
| 1.3 | 22 NOV 2018 | PPD | Based on client comments |
| 2.0 | 26 NOV 2018 | PPD | Final Version |
| 2.0 | 04 FEB 2019 | PPD | Final Version |
| 2.0 | 04 FEB 2019 | PPD | Based on client comments |
| 2.0 | 13 FEB 2019 | PPD | Final Version |

## 5. Purpose of the Statistical Analysis Plan

The purpose of this Statistical Analysis Plan (SAP) is to document technical and detailed specifications for the final analysis of data collected for protocol EMR200505\_506. Results of the analyses described in this SAP will be included in the Clinical Trial Report (CTR). Any post-hoc, or unplanned analyses performed to provide results for inclusion in the CTR but not identified in this prospective SAP will be clearly identified in the CTR.

The SAP is based upon trial protocol and protocol amendments and is prepared in compliance with International Council for Harmonization of Technical Requirements for Pharmaceuticals for Human Use (ICH) E9 Guidelines. The SAP focused on the improvement of microvascular function by positron emission tomography (PET) after twelve-week treatment of oral nicorandil in female non obstructive CAD patients. Statistical analyses for other variables such as the improve of myocardial blood flow (MBF) by rest and stress PET, the improve of heart function by echocardiography, the improve of angina attacks after twelve-week treatment of oral nicorandil and safety variables are also added in this version of SAP.



# 6. Summary of Clinical Trial Features

| Study Title | An interventional, pilot study to evaluate the efficacy of |
|---|---|
| | oral nicorandil on improving microvascular function in |
| | female non obstructive CAD patients (SPET study) |
| Study number | EMR200505_506 |
| Study Phase | IV |
| Study Center(s)/Country(ies) | 1 (hospital)/1 (country) |
| Study Background | Quantification of myocardial blood flow (MBF) and |
| | MFR has incremental values in the evaluation of the |
| | prognosis for patients with cardiovascular disease. There |
| | has been significant variation in the diagnostic criteria |
| | used to define CMD. The current gold standards for |
| | clinically assessing microvascular function have been |
| | CFR using invasive testing and positron emission |
| | tomography (PET). A CFR<2.0 strongly suggests |
| | coronary microvascular disease, and related to patients |
| | CV outcomes. However, many treatment studies have |
| | included subjects with CFR values >3 in their analysis. |
| | This study use a CFR<3.0 as a cutoff value for judging |
| | whether patient has coronary microvascular decease. |
| | Nicorandil is a unique dual pharmacological mechanism |
| | anti-anginal agent with adenosine triphosphate sensitive |
| | potassium (K <sub>ATP</sub> ) channel agonist and nitrate-like |
| | properties. It opens $K_{ATP}$ channels in the vascular |
| | smooth muscle cell, leading to K <sup>+</sup> efflux and membrane |
| | hyperpolarization, which in turn reduces Ca <sup>2+</sup> influx, |
| | including closing voltage-sensitive calcium channels |
| | (VOC). Its K <sub>ATP</sub> channel opening effect also inhibits |
| | Ca <sup>2+</sup> release from the sarcoplasmic membrane. The |
| | concentration of intracellular free Ca <sup>2+</sup> then decreases. |

| | Arterial vasodilation is therefore predominant. $K_{ATP}$ |
|---|---|
| | _ |
| | channel is one of the most critical target spots that |
| | regulates the tone of coronary arterioles (with diameter |
| | <200 μm) |
| Study objectives | Primary objective: |
| | To avaluate the improvement of microvescular function |
| | To evaluate the improvement of microvascular function |
| | by positron emission tomography (PET) after twelve- |
| | week treatment of oral nicorandil in female non |
| | obstructive CAD patients; |
| | Secondary objectives: |
| | To evaluate the improve of myocardial blood flow |
| | (MBF) by rest and stress PET after twelve-week |
| | treatment of oral nicorandil |
| | • To evaluate the improve of heart function by |
| | echocardiography after twelve-week treatment of |
| | oral nicorandil |
| | To evaluate the improve of angina attacks after |
| | twelve-week treatment of oral nicorandil |
| Primary endpoint(s) | Comparison of myocardial blood flow reserve (MFR) |
| | between baseline and after twelve-week treatment |
| Secondary endpoint(s) | Comparison of below items between baseline and after |
| | twelve-week treatment |
| | <ul> <li>MBF by rest and stress PET</li> </ul> |
| | • Parameters of heart function by Echocardiography: |
| | o Cardiac systolic function: Ejection Fraction |
| | (EF%), left ventricular end-systolic dimension |
| | (LVESD), left ventricular wall thickness |
| | Cardiac diastolic function: E/A ratio |
| | Seattle Angina Questionnaire (SAQ) score |
| | South Ingina Questionian (SIIQ) soole |

| Study Design | This is a single-center, interventional, pilot clinical trial. |
|---|---|
| | 11-20 patients will be enrolled in the treatment group |
| | who will take oral Nicorandil 5mg, t.i.d for 12 weeks. |
| | For all the patients, rest cardiac PET and stress cardiac |
| | • |
| | PET will be tested at both screening period and end of |
| | study. Other laboratory parameters and clinical |
| | symptoms will be collected at baseline, 4 weeks, 8 |
| | weeks and 12 weeks of treatment. There will be 5 visits |
| | from the beginning to the end of the study |
| Planned number of subjects | 11-20 |
| Schedule of visits and assessments | Screening visit: ECG, lab tests, MFR by rest and stress |
| | PET, UCG; |
| | Visit 1 (week 0): ECG, SAQ; |
| | Visit 2 (week 4): ECG; |
| | Visit 3 (week 8): ECG; |
| | Visit 4 (week 12): ECG, lab tests, MFR by rest and |
| | stress PET, UCG |
| Eligibility Criteria | Inclusion criteria: |
| | Female |
| | Patients aged 18-70 years |
| | • Patients with typical stable angina but without |
| | coronary obstruction (defined as coronary occlusion |
| | < 50%) by invasive coronary angiography or |
| | coronary computed tomography angiography (CTA) |
| | in recent three months |
| | • All other long acting cardiovascular disease |
| | medicines, including but not limited to |
| | aspirin/clopidogrel, CCB, ACEI/ARB, $\beta$ -blockers, |
| | statins, ivabradine, trimetazidine, et al, should be |

## period

For patients who met these four criteria above, MFR will be tested by stress PET. Patients whose MFR
 <3.0 could be included in the study</li>

#### **Exclusion criteria:**

- Severe or uncontrolled hypertension (resting SBP ≥ 160 mmHg, or resting DBP ≥ 100 mmHg at screening period)
- Patients with shock (including cardiogenic shock), or hypovolemia
- Severe hypotension (resting SBP < 90 mmHg, or resting DBP < 60 mmHg)</li>
- Significant valvular heart disease, congenital heart disease or cardiomyopathy
- Congestive heart failure (NYHA III-IV), echocardiographic ejection fraction < 45%
- Acute pulmonary edema
- Hepatic or renal dysfunction, defined as:
  - Serum Alanine Aminotransferase (ALT) > triple
     of the normal value upper limit;
  - Serum Aspartate Aminotransferase (AST) >
     triple of the normal value upper limit
  - Serum creatinine > twice of the normal value upper limit
- Glaucoma
- Active peptic ulcer or active skin ulcer
- Taking glyburide, PDE-5 inhibitors, soluble guanylate cyclase stimulator(s)
- Known to be hypersensitivity to nicorandil, nitrates, niacin, or any of the excipient



| | With contraindication to complete stress PET test |
|---|---|
| | No legal ability and legal ability is limited |
| | • Patients unlikely to cooperate in the study or with |
| | inability or unwillingness to give informed consent |
| | Child-bearing period women without effective |
| | contraceptive measures, pregnancy and lactation |
| | Participation in another clinical trial within the past |
| | 30 days |
| | • Other significant disease that in the Investigator's |
| | opinion would exclude the subject from the trial |
| Investigational Medicinal Product (s): | Nicorandil (SIGMART® Tablets 5.0 mg) / Oral / t.i.d, |
| dose/mode of administration/ dosing | g 12 weeks |
| schedule | |
| Reference therapy(ies): dose/mode of | Patients have already received the current standard |
| administration/dosing schedule | therapy strategy, if conditions permitted, |
| | aspirin/clopidogrel, ACEI/ARB, $\beta$ -blockers, CCBs, and |
| | statins should be included; |
| | All the medicines mentioned above and other anti- |
| | angina medicines (except nitroglycerine) need to be |
| | stabilized at least two weeks before screening period; |
| | All subjects will start taking nicorandil after enrollment. |



# Schematic diagram of the study plan:



# **Schedule of Assessments**

| | Screening visit | Visit 1 | Visit 2 | Visit 3 | Visit 4 |
|---|---|---|---|---|---|
| | (Day -14 to 0) | (Day 1±3) | (Day 28±3) | (Day 56±3) | (Day 84±3) |
| Signing the ICF | X | | | | |
| Demographic data | X | | | | |
| Inclusion and exclusion criteria | X | | | | |
| Medical history | X | | | | |
| Body weight and height | X | | | | X |
| Waist circumference | X | | | | X |
| Vital signs | X | X | X | X | X |
| Physical examination | X | X | X | X | X |
| ECG | X | X | X | X | X |
| Full blood count | X | | | | X |
| Hepatic and renal functions | X | | | | X |
| Blood glucose and lipids | X | | | | X |
| Echocardiography | X | | | | X |
| Rest and stress PET | X | | | | X |
| SAQ | | X | | | X |
| Cardiovascular events | | X | X | X | X |
| Sigmart® therapy (For treatment group only) | | X | X | X | X |
| Adverse event record | X | X | X | X | X |
| Medication possession ratio (MPR) | X | | | | X |
| Concomitant medicine | X | X | X | X | X |



## 7. Sample Size

The null hypothesis is that there is no difference between MFR at baseline and MFR after twelve weeks treatment. The alternative hypothesis is that the MFR after twelve weeks treatment is higher than the MFR at baseline.

Suppose the difference of MFR follows normal distribution, and the following assumptions are made to determine the sample size:

- The mean value of difference of MFR is 0.55
- The standard deviation of difference of MFR is 0.56
- Alpha = 0.05 (two sided)
- Power = 0.80

A sample size of 11 patients will be required to reach this goal. Assuming a drop-out rate of 30%, then a total of 15 patients will be recruited into this study. According to the recruitment progress, if there have been 11 patients complete their follow-up period, this study could be accomplished when meet the end of the anticipated period of the whole study.

## 8. Overview of Planned Analyses

This SAP describes final analysis of the study. No interim analyses are planned for this study.

## 9. Changes to the Planned Analyses in the Observational Study Protocol

The statistical methods as described in the protocol were adopted.

## 10. Analysis Sets

## **Screening Population**

The screening population will include all subjects who provide written informed consent and who undergo screening assessments, regardless of treatment status in the trial.



## **Intention-to-treat (ITT) Population**

The ITT population is the subset of screening population, and it should include all subjects who receive at least one dose of trial treatment.

## Per Protocol (PP) Population

The PP population will be the subset of the ITT population that is compliant with the protocol and characterized by criteria such as:

- 1) Measurement of the primary endpoint both at baseline and after twelve week treatment.
- 2) Absence of any major protocol deviation.

The PP population will be identified before database lock and will be used to test the primary endpoint. It will be considered a secondary population.

## **Safety Population**

The safety population will include all subjects who received at least one dose of trial treatment.

The ITT population will be used primarily to present baseline characteristics and analyze efficacy data. Selected efficacy analyses will be repeated for the PP population. The safety population will be used to summarize the safety data.

#### 11. General Specifications for Statistical Analyses

Statistical analysis will be made utilizing Statistical Analysis System (SAS) version 9.1.3 or higher.

Descriptive statistics such as

- Number of subjects (n), number of subjects with missing values (Missing),
- Mean, Standard Deviation (SD),
- Median, First Quartile (Q1), Third Quartile (Q3),
- Minimum and Maximum

will be provided for all continuous variables.



Mean, Median, Q1 and Q3 will have more than one decimal place than the raw data and SD will have 2 decimal places more than the raw data. The decimal place for minimum and maximum values will be same as the raw data.

The frequency (n) and percentage (%) will be calculated for all categorical variables including missing observations and the percentages will be rounded off to one decimal place.

95% Confidence Interval (CI) will be provided wherever applicable.

If day is missing for any date variable then it will be replaced by 1<sup>st</sup> day of the month. Similarly, missing month will be replaced by 1<sup>st</sup> month of the year.

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 21.0 or higher terminology for System Organ Class (SOC) and Preferred Term (PT).

#### Handling of missing data

Missing information will be captured for quantitative as well as qualitative variables by the category "Missing" in the summary statistics. If there are no missing values this will be indicated by "0". Unless otherwise specified missing data will not be replaced.

## 12. Trial Subjects

## 12.1 Disposition of Subjects and Discontinuations

A table with

- Number of subjects screened
- Number of screen failure subjects
- Number of subjects enrolled in the study
- Number of subjects in ITT population
- Number of subjects in PP population
- Number of subjects in safety population
- Number of subjects (ITT population) who completed the study



 Number of subjects (ITT population) who discontinued from the study together with primary reason for study discontinuation (Adverse event/ Lost to follow-up/ Lack of efficacy/ Death/ Withdrew Consent/ Study reached predefined end/ Other)

will be summarized as number and percentage.

#### 12.2 Outliers

Listing will be provided for subjects with outliers (if data available). Extreme data that are not explainable from clinical point of view are considered as outliers. Subjects with such outliers will be identified before the database lock. These outlier data will not be included in the analysis.

## 13. Demographics and Other Baseline Characteristics

### 13.1 Demographics

The quantitative variable

• Age (years)

will be summarized by descriptive statistics from ITT Population.

The age variable will be calculated by using below formula:

Age (years) = (Date of Informed consent - Date of Birth) + 1

If day is missing for any date variable then it will be replaced by 1<sup>st</sup> day of the month. Similarly, missing month will be replaced by 1<sup>st</sup> month of the year.

The qualitative variables

- Sex (Female)
- Race (Asian/ Other)

will be summarized as number and percentage from ITT Population.



## 13.2 Medical History

The following information will be collected for the medical history of the subjects:

## History of Hypertension/Heart Failure/Diabetes

Listing will be provided for History of Hypertension/Heart Failure/Diabetes for ITT Population.

## **Other Medical History**

Listing will be provided for history of any other medical conditions for ITT Population.

## **History of Angina Pectoris**

The quantitative variables

- Duration of Angina Pectoris (Years)
- Frequency of angina attacks in recent one month per week

will be summarized by descriptive statistics from ITT Population.

The qualitative variable

• Classification (Stable/ Unstable)

will be summarized as number and percentage from ITT Population.

## 14. Previous or Concomitant Medications/Procedures

Listings will be provided for Prior and Concomitant Medications and Concomitant Procedures for all individual subjects for ITT Population.



## 15. Treatment Compliance and Exposure

## **Treatment Compliance**

The quantitative variables

- Number of tablets to be taken
- Number of tablets taken
- Percentage (%)

will be summarized using descriptive statistics from Safety Population.

The qualitative variable

• Compliance (Good (80%-100%) / Insufficient (<80% or >100%))

will be summarized as number and percentage from Safety Population.

# SIGMART® Administration

The quantitative variables

- Total duration of Sigmart® administration (Days)
- Total dose of Sigmart<sup>®</sup> administration (mg)

will be summarized using descriptive statistics from Safety Population.

Total duration of Sigmart<sup>®</sup> administration will be calculated by using below formula:

Total duration Sigmart<sup>®</sup> Administration (Days) = (Last dose of SIGMART<sup>®</sup> Administration End date – First dose of SIGMART<sup>®</sup> Administration Start date) + 1.

Total dose (mg) of Sigmart<sup>®</sup> administration will be calculated by using below formula:

Total dose (mg) of Sigmart<sup>®</sup> Administration = Sum of (Daily dose of Sigmart<sup>®</sup> Administration \* number of treatment days for the dose).



The qualitative variables

- Change in dose (No change/ Dose adjusted/ No dose)
- Reason for dose adjustment (Adverse event/ Titration/ Other)
- Reason for no dose (Adverse event/ Missed dose/ Other)

will be summarized as number and percentage from Safety Population.

## 16. Endpoint Evaluation

## 16.1 Primary Endpoint Analyses

The primary endpoint is comparison of myocardial blood flow reserve (MFR) between baseline and after twelve-week treatment. The null hypothesis is that there is no difference between MFR at baseline and MFR after twelve week treatment. The alternative hypothesis is that the MFR after twelve week treatment is higher.

The quantitative variable

• Myocardial blood flow reserve (MFR)

will be summarized using descriptive statistics at baseline, visit 4 (week 12) and change from baseline from ITT and PP populations. Two-sided 95% confidence interval (CI) will be calculated for the difference between MFR at baseline and after twelve week treatment.

Paired T-test or Wilcoxon Signed Rank test will be used to compare the myocardial blood flow reserve (MFR) between baseline and after twelve-week treatment based on the normality assumption of the data.



## 16.2 Secondary Endpoint Analyses

## MBF by rest and stress PET

The quantitative variables

- Rest PET-MBF (ml/gm/min)
- Stress PET-MBF (ml/gm/min)

will be summarized using descriptive statistics at baseline, visit 4 (week 12) and change from baseline from ITT and PP populations. The same analysis as mentioned for primary endpoint (MFR) will be performed for MBF by rest and stress PET.

## **Echocardiography**

The quantitative variables

- Ejection Fraction (EF) (%)
- Left ventricular end systolic dimension (LVESD) (mm)
- Interventricular septum thickness (IVST) (mm)
- Left ventricular posterior wall thickness (PWT) (mm)
- E/A Ratio

will be summarized using descriptive statistics at baseline, visit 4 (week 12) and change from baseline from ITT and PP populations. The same analysis as mentioned for primary endpoint (MFR) will be performed for all Echocardiography variables.

#### Seattle angina questionnaire (SAQ)

The Seattle angina questionnaire (SAQ) score will be classified into five dimensions: physical limitation (question 1), anginal stability (question 2), anginal frequency (question 3-4), treatment satisfaction (question 5-8) and disease perception (question 9-11). The sum of score in each

dimension will be calculated respectively, and then transformed into the standard score between 0 and 100:

(Sum of Score - the minimum value of score in this dimension) X 100 (The range of score in this dimension)

For example: Suppose the sum of score in dimension 1 is 43, and the minimum and maximum of score in this dimension is 1 x 9=9 and 6 x 9=54 respectively. So the standard score in this dimension is  $\frac{43-9}{54-9} \times 100 = 75.55$ ;

Suppose the sum of score in dimension 2 is 2 and the minimum and maximum of score in this dimension is 1 and 5 respectively. So the standard score in this dimension is  $\frac{2-1}{5-1} \times 100 = 25$ 

The scores for the following dimensions

- Physical limitation
- Anginal stability
- Anginal frequency
- Treatment satisfaction
- Disease perception

will be summarized using descriptive statistics at visit 1 (week 0), visit 4 (week 12) and change from visit 1 (week 0) from ITT and PP populations. The same analysis as mentioned for primary endpoint (MFR) will be performed for each dimension.

## 17. Safety Evaluation

Safety evaluation includes the summary of safety endpoints such as AEs, TEAEs, SAEs, laboratory tests, ECG parameters and vital signs during the study based on safety population.

## 17.1 Adverse Reactions / Events

AEs will be summarized per subject using number and percentage by SOC and PT from Safety Population. If an AE is reported for a subject more than once during treatment, the worst severity and the worst relationship to trial treatment will be tabulated. Listings will also be provided for all the AEs.

AEs will be coded using MedDRA version 21.0 or above.

#### 17.1.1 All Adverse Events

All AEs and Treatment Emergent Adverse Events (TEAE) will be summarized using number and percentage by MedDRA-SOC and PT within SOC for severity, relationship, causality factors other than study treatment, action taken with study medication and outcome. The AEs and TEAEs reported under the category "Related" will be considered as treatment-related AEs and TEAEs. Missing will also be considered as related to the treatment. PT within SOC and primary SOC will be given in alphabetical order from safety population.

**TEAE period:** Occurrence of AE in nicorandil period, which means from day 0 to last visit.

#### 17.1.2 Adverse Events Leading to Trial or Treatment Discontinuation

AEs leading to study termination will be summarized by MedDRA-SOC and PT within SOC.

## 17.2 Deaths, Other Serious Adverse Events, and Other Significant Adverse Events

#### **17.2.1** Deaths

If any death is reported it will be presented as case narrative.

Listings will also be provided.

#### 17.2.2 Serious Adverse Events

Serious adverse events (SAEs) will be summarized per subject using number and percentage by SOC and PT from safety population.



All SAEs will be summarized using number and percentage by MedDRA-SOC and PT within SOC for severity, relationship, causality factors other than study treatment, action taken with study medication and outcome. The SAEs reported under the category "Related" will be considered as treatment-related SAEs. Missing will also be considered as related to the treatment. PT within SOC and primary SOC will be given in alphabetical order from safety population.

#### 17.3 Clinical Laboratory Evaluation

#### Hematology

The quantitative variables

- Hemoglobin (HGB) (g/dL)
- Erythrocytes (RBC) (10^9/L)
- White blood cells (WBC) (K/ul)
- Neutrophils (NEUT) (10^3/mcL)
- Platelet count (PLAT) (10^3/mcL)

will be summarized using descriptive statistics including standard error of mean (SEM) and 95% confidence interval at baseline, visit 4 (week 12) and change from baseline from Safety Population.

Unit conversion for Hematology will be done at the time of analysis appropriately.

#### **Bio Chemistry**

The quantitative variables

- Alanine Aminotransferase (ALT) (IU/L)
- Aspartate aminotransferase (AST) (IU/L)
- Blood Urea Nitrogen (BUN) (mg/dL)
- Creatinine (CREAT) (mg/dL)
- Total Cholesterol (mmol/L)



- Triglycerides (µmol/l)
- HDL cholesterol (µmol/l)
- LDL Cholesterol (µmol/l)
- Potassium (mEq/L)
- Sodium (mEq/L)
- Myocardial Enzymes (CKMB) (IU/L)

will be summarized using descriptive statistics including standard error of mean (SEM) and 95% confidence interval at baseline, visit 4 (week 12) and change from baseline from Safety Population.

Unit conversion for Bio Chemistry will be done at the time of analysis appropriately.

## **Routine Urine Test (Urinalysis)**

The quantitative variables

- pH
- Specific gravity

will be summarized using descriptive statistics including standard error of mean (SEM) and 95% confidence interval at baseline, visit 4 (week 12) and change from baseline from Safety Population.

Shift tables for below mentioned qualitative Routine Urine Test (Urinalysis) variables will be summarized with number and percentage of change among the results Normal, Trace/+, ++, +++ & ++++ at Baseline and Visit 4 (Week 12) from safety population.

- Protein
- Glucose
- Ketone
- Nitrite



- Leukocytes
- Hemoglobin
- Red blood cells
- Bilirubin

#### **Other Lab Tests**

The quantitative variable

Fasting Blood Glucose (µmol/l)

will be summarized using descriptive statistics including standard error of mean (SEM) and 95% confidence interval at baseline, visit 4 (week 12) and change from baseline from Safety Population.

Unit conversion for Fasting Blood Glucose will be done at the time of analysis appropriately Shift tables for below mentioned qualitative Other Lab Tests variables will be summarized with number and percentage of change among the results Positive and Negative at Baseline and Visit 4 (Week 12) from safety population.

• Urine Pregnancy Test (Positive / Negative)

Listings will also be provided for all the Clinical Laboratory parameters.

### 17.4 Electrocardiogram (ECG)

The quantitative variable

• Heart Rate (beats/min)

will be summarized using descriptive statistics including standard error of mean (SEM) and 95% confidence interval at baseline, visit 4 (week 12) and change from baseline from Safety Population.



The qualitative variables

- Rhythm (Sinus rhythm/ Arrhythmia)
- Cardiac hypertrophy (Yes/No)
- ST-T Change (Abnormal) (Yes/No)

will be summarized as number and percentage at all available visits from Safety Population. Listings will also be provided for ECG Parameters.

#### **Vital Signs**

The quantitative variables

- Systolic Blood pressure in Sitting Position (mmHg)
- Diastolic Blood pressure in Sitting Position (mmHg)
- Resting Heart rate (beats/minute)
- Height (cm)
- Weight (kg)
- BMI (kg/m<sup>2</sup>) (Auto calculated in database)
- Waist circumference (cm)

will be summarized using descriptive statistics including standard error of mean (SEM) and 95% confidence interval at all available visits and change from baseline from Safety Population.

Conversion formula for Waist circumference: cm = inches \* 2.54.

Listings will also be provided for Vital Signs Parameters.

## 17.5 Physical Examination

All abnormalities occurring or worsening in physical examination after putting signature in the informed consent will be recorded in the Adverse Events section unless otherwise stated by the protocol. Hence, physical examination parameters will not be summarized separately.



## 18. Benefit risk assessment

Not applicable.

## 19. References

- 1. Protocol Number: EMR200505\_506, Dated 15 APR 2018, Protocol Amendment <III>
- 2. Case Report Form Version 4.0 dated 23 JAN 2019
- 3. ICH E3 "Structure and Content of Clinical Study report" and E9- "Statistical Principles for Clinical Trials".

## 20. Appendices

Not applicable.

